CLINICAL TRIAL: NCT00181623
Title: Recombinant Human Prolactin for Lactation Induction in Prolactin Deficient Mothers
Brief Title: Recombinant Human Prolactin for Lactation Induction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Corrine Welt, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003P001209-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2013-05-09 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Lactation
Keywords: Lactation; Breastfeeding; Prolactin; Primary lactation insufficiency
MeSH Terms: conditions — Breast Feeding

ARMS (1):
- recombinant human prolactin treatment (Experimental): Open label twice daily recombinant human prolactin
  Interventions: Drug: Recombinant Human Prolactin

INTERVENTIONS:
Drug: Recombinant Human Prolactin

SUMMARY:
The purpose of the study is to assess the safety and determine the effects of the hormone prolactin on lactation (breast milk production).

DETAILED DESCRIPTION:
The efficacy of recombinant human prolactin (r-hPRL) for treatment of primary lactation insufficiency in women with prolactin deficiency, either congenital or acquired, will be examined. Subjects will participate in an open-label study of r-hPRL administration for prolactin deficiency. On study day 1, subjects will be seen between 8 and 10 am. A baseline prolactin level will be obtained. Subjects will subsequently be taught to use a breast pump by a designated lactation consultant and will pump for 10 minutes at each breast, simultaneously or sequentially. Any milk production will be recorded, along with milk volume throughout the study. Prolactin levels will be obtained every 10 minutes for 60 minutes after pumping begins, then every 30 minutes for a total of 3 hours. At 3 hours, r-hPRL 60 mg/kg will be administered SC. Blood will be drawn every 2 hours for 8 hours to obtain a peak prolactin level. Vital signs will be monitored every 15 minutes for the first hour, then every 2 hours for a total of 8 hours. Subjects will again pump both breasts 0, 3 and 6 hours after the r-hPRL injection, to maintain an every 3 hour schedule. Any milk production will be recorded. Subjects will administer their second dose of SC r-hPRL 12 hours after the first dose.

Subjects will continue every 12 hour SC r-hPRL administration for the next 28 days. They will also pump every 3 hours, with the exception of a 5 hour break for sleep at one time during the 24 hours, as long as the total number of pumping episodes equals 8. Subjects will record any milk production and will call as soon as any milk is expressed. When the first milk is produced, the infant will not be allowed to suckle at the breast until the milk is tested and readministered to the infant in a controlled setting to avoid any potential risks or r-hPRL exposure to the infant in the interim. After each pumping episode, if no milk is produced mothers will be encouraged to let their infants feed at the breast using a Lact-Aid device.

Subjects will be seen in the GCRC, weekly for 28 days. At each visit, subjects will have a breast exam for galactorrhea and a baseline prolactin level, then subjects will administer their own SC r-hPRL injection and pump at 0, 3 and 6 hours after r-hPRL administration, as described above. Any milk production will be recorded. In addition, at the end of week 1 and on the final day, r-hPRL will be administered, blood will be drawn every 2 hours for prolactin levels as on the first day of the injection, for a total of 8 hours, and subjects will pump and milk volume will be recorded at 0, 3 and 6 hours after r-hPRL administration.

When at least 0.25 cc of milk is produced by pumping, it will be sent for a prolactin level measurement to determine whether levels are elevated compared to levels in the control milk. If the prolactin level is not elevated, milk will be readministered to the infant. When breast milk is first given to the infants, they will be monitored in the GCRC under the supervision of a neonatologist, with vital signs, including temperature, measured every hour after feeding for 4 hours. The mother will also record stool and gastric output and any changes noted in the quality or quantity of output for the following 24 hours. If any significant and adverse changes in vital signs or gastric output are observed, any additional stored breast milk will be discarded and the study stopped. After the prolactin level in milk has been documented in the normal range and milk readministered to the infant under supervision in the GCRC, mothers will continue to pump immediately after the am r-hPRL dose, but at all other times will be encouraged to breastfeed.

When at least 1 cc of milk is available, milk composition will also be analyzed for fat, protein, glucose, lactose and IgA levels (see Procedure for Analyzing Collected Milk, above). Studies in mothers of premature infants will be performed before starting this protocol. If the level of any of these components is 50% below the lower limit of normal, breast milk will be supplemented with formula at a ratio determined by the neonatologist to ensure that all nutrients are received.

After completing 28 days of every 12 hour r-hPRL administration, breast milk production will continue to be monitored for a 14 day control period. Subjects will be seen at 7 and 14 days after their final prolactin injection. After a baseline prolactin level is drawn, milk will be pumped until the breasts are emptied. Blood will be drawn at baseline and then every 10 minutes for 60 minutes, then every 30 minutes for a total of 3 hours to obtain a prolactin peak.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, aged 18-45 years
* Prolactin deficiency due to congenital deficiency, surgery or radiation, or Sheehan's syndrome during the current or previous pregnancies, for women who desire to breastfeed their infants.
* Postpartum at the time of study participation
* Milk must fail to come in by 2-4 days after delivery.
* Prolactin levels will be less than the lower limit of normal for the assay performed. If a subject is postpartum, prolactin levels will be less than the normal range for postpartum women (<= 138.0 ± 11.9 ng/mL).
* Free T4 index must be normal either on or off thyroid hormone replacement.
* Fasting am cortisol or 1 hour Cortrosyn 0.25 mg stimulated cortisol must be normal (>18 mg/dL). If it is not normal, subjects must be on glucocorticoid replacement and have no symptoms of adrenal insufficiency.
* History of normal spontaneous puberty or Tanner stage V breast development after previous estrogen replacement therapy.

Exclusion Criteria:

* Current use of medications known to increase or decrease prolactin
* Anatomical breast abnormalities
* Previous mammoplasty
* Breast augmentation
* Current use of hormonal contraception
* Allergies to mannitol
* Medications contraindicated for breastfeeding mothers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2005-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine K Welt, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Iwama S, Welt CK, Romero CJ, Radovick S, Caturegli P. Isolated prolactin deficiency associated with serum autoantibodies against prolactin-secreting cells. J Clin Endocrinol Metab. 2013 Oct;98(10):3920-5. doi: 10.1210/jc.2013-2411. Epub 2013 Aug 12. PMID 23940128
- [Derived] Powe CE, Puopolo KM, Newburg DS, Lonnerdal B, Chen C, Allen M, Merewood A, Worden S, Welt CK. Effects of recombinant human prolactin on breast milk composition. Pediatrics. 2011 Feb;127(2):e359-66. doi: 10.1542/peds.2010-1627. Epub 2011 Jan 24. PMID 21262884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2005-2008 Academic Hospital, clinical research center
Groups:
- Recombinant Human Prolactin Treatment: Open label twice daily recombinant human prolactin 60 mcg/kg
  Recombinant Human Prolactin :
Period: Overall Study
Arm/Group | Recombinant Human Prolactin Treatment
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Recombinant Human Prolactin Treatment: Open label twice daily recombinant human prolactin
  Recombinant Human Prolactin :
Arm/Group | Recombinant Human Prolactin Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Breast Milk Production
Description: Treatment group
Time Frame: 28 days
Population: One subject did not qualify after screening.
Measure: Mean (Standard Error); unit: mL/day
Arm/Group | Recombinant Human Prolactin Treatment
Number analyzed (Participants) | 5
mL/day | 66.1 (8.3)

2. Secondary Outcome: Breast Milk Prolactin Levels
Description: Treatment group
Time Frame: 28 days
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | Recombinant Human Prolactin Treatment
Number analyzed (Participants) | 5
mcg/L | 118 (25)

ADVERSE EVENTS:
Arm/Group | Recombinant Human Prolactin Treatment
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Prolactin Treatment (N=5)
Tingling in hands (Nervous system disorders) | 1 (1)
Red marks at injection site (Skin and subcutaneous tissue disorders) | 1 (1)
Tiredness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small numbers as this was an orphan disease trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes